CLINICAL TRIAL: NCT03624751
Title: Follow up for Patients With Thyroid Cancer Planed for Radioiodine Scan or Treatment
Status: Recruiting | Type: Observational
Sponsor: Taichung Veterans General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CE18104A
Record Dates: First submitted 2018-05-24; First posted 2018-08-10 (Actual); Last update posted 2018-08-10 (Actual); Status verified 2018-08

CONDITIONS: Thyroid Cancer
MeSH Terms: conditions — Thyroid Neoplasms | interventions — Iodine-131

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: radioiodine — Patients with thyroid cancer need to choose between Thyrogen® injection and Eltroxin® withdrawal before radioiodine therapy or scan.

SUMMARY:
The prevalence of thyroid cancer has increased in recent decades. Patients with thyroid cancer need to choose between Thyrogen® injection and Eltroxin® withdrawal before radioiodine therapy or scan. This is a prospective, observational study, aiming to observe the difference of metabolic profiles between patients choose Thyrogen® injection and Eltroxin® withdrawal.

DETAILED DESCRIPTION:
1. Objective： To observe the difference between Thyogen® injection or Eltroxin® withdrawal on metabolic profile.
2. Background and method:： The prevalence of thyroid cancer has increased in recent decades. Patients with thyroid cancer need to choose between Thyrogen® injection and Eltroxin® withdrawal before radioiodine therapy or scan. This is a prospective, observational study, aiming to observe the difference of metabolic profiles between patients choose Thyrogen® injection and Eltroxin® withdrawal.

Inclusion ： Patient number: 500人

Inclusion criteria :

1. Patients with diagnosis of thyroid cancer。
2. Patients who need radioiodine therapy or scan。

Exclusion criteria:

1. Patients cannot cooperate with blood test.。
2. Patients cannot cooperate with radioiodine therapy。 Study design： Prospective, observational study。

Method： We will collect 20cc blood and 20 cc urine before and after radioiodine therapy during each visit (total 3 visits) and check lipid profiles, glucose profiles and inflammation markers. We will compare the difference between results of patients undergoing Thyrogen® injection and Eltroxin® withdrawal.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with diagnosis of thyroid cancer。
2. Patients who need radioiodine therapy or scan。

Exclusion Criteria:

1. Patients cannot cooperate with blood test.。
2. Patients cannot cooperate with radioiodine therapy。

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with diagnosis of thyroid cancer
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2018-06-30 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
Zung's Self-reported depression scale | 1 month
  Depression symtpoms

SECONDARY OUTCOMES:
Brain-derived neurotrophic factor | 1 month
  BDNF
orexin | 1 month
  An associated factor for depression
Body composition | 1 months
  Fat component percentage to lean mass percentage ratio
VCAM-1 | 1 months
  adhesion molecules
CRP | 1 months
  inflammation marker
Metabolic syndrome | 1 months
  The number of conponents for metabolic syndrome

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Endocrinology and Metabolism in Taichung Veterans General Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided